CLINICAL TRIAL: NCT03340428
Title: Corrections2Community: Post-release Retention in HIV Care for Ex-inmates in South Africa
Brief Title: Post-release Retention in HIV Care for Ex-inmates in South Africa
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Aurum Institute (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: IRB00181117; 1R34MH115777 (NIH)
Record Dates: First submitted 2017-11-08; First posted 2017-11-13 (Actual); Results first posted 2021-04-27 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2021-03

CONDITIONS: Hiv; Adherence, Patient
Keywords: incarceration; linkage to care; retention in care
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Patient Compliance

STUDY DESIGN:
Intervention Model Description: Individually randomized trial with 2:1 allocation to the intervention compared to care as usual
Who Masked: Investigator, Outcomes Assessor
Masking Description: Intervention arm will be masked to the field researchers and the investigators until unblinding during final analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transition Community Adherence Club (TCAC) (Experimental): Participants in this arm will be referred to join a facilitated group setting for HIV on release from incarceration. This arm will provide HIV care services in a facilitated group setting to provide medical and psychosocial needs of participants.
  Interventions: Behavioral: Transition Community Adherence Club (TCAC)
- Care as usual (CAU) (No Intervention): Care as usual participants will be referred to routine clinic HIV care on release from corrections.

INTERVENTIONS:
Behavioral: Transition Community Adherence Club (TCAC) — A behavioral intervention targeting stigma and care challenges through care delivery, social capital through a group setting, improved job prospects through referrals and training, and substance use through referrals. Participants assigned to this group will meet at least every month in a group of 5-15 members for approximately 2 hours. During the meeting there will be facilitated group discussion, an interactive curriculum including life skills, economic skills, HIV and health, and disclosure and stigma. Individual health screening and distribution of prepackaged medications conclude the session. Individual referrals for specific services (e.g. mental health or substance use management) will be available.
  Other Names: Transition Community Adherence Club
  Arms: Transition Community Adherence Club (TCAC)

SUMMARY:
HIV remains the leading cause of death in South Africa as a result of a failure of people living with HIV to seek HIV treatment and be retained in care. After initiating antiretroviral therapy while incarcerated, most ex-inmates fail to remain engaged in care. The goal of this research is to reduce mortality, morbidity, and HIV transmission by developing an actionable approach to retaining these individuals in HIV care.

DETAILED DESCRIPTION:
To pilot a randomized clinical trial (RCT) of a transition adherence club (TCAC) versus traditional care, among ex-inmates receiving antiretroviral therapy in South Africa, to study feasibility, acceptability, and preliminary effectiveness using mixed methods.

Investigators will pilot an RCT of the TCAC compared to traditional care among inmates/ex-inmates measuring transition in care, six-month viral load suppression, and follow-up of participants. Feasibility will be assessed by process measures. Acceptability will be assessed using in-depth interviews among 36 participants and 10 staff. Effectiveness will be assessed by a difference in proportions in-care with an undetectable viral load at 6 months and difference in bonding social capital and care satisfaction between arms.

ELIGIBILITY:
Inclusion Criteria:

* Currently incarcerated (either an offender/sentenced inmates or awaiting trial inmate/remandee)
* Housed at one of the study correctional facilities (including participating satellite centres)
* Diagnosed with HIV
* Currently receiving antiretroviral therapy
* Anticipated release or trial date within 3 months of study enrollment
* Self-report expected to reside within Ekurhuleni, Tshwane, or Johannesburg districts of Gauteng Province and within proximity to one of the TCAC sites (within 20 km, 45 minute travel time, or two local taxi minibus rides)
* Agree to post-discharge follow-up
* Medically stable based on DCS health assessment (including not pregnant)
* On antiretroviral therapy (ART) for >3 months at the expected time of corrections release

Exclusion Criteria:

* Failure to provide informed consent to be followed up by study staff after release
* Unable to speak one of the study languages (English, Sesotho, isiXhosa, isiZulu, Setswana, Xitsonga, and Afrikaans)

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 176 (Actual)
Dates: Start 2019-03-09 (Actual); Primary Completion 2020-08-01 (Actual); Study Completion 2020-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Hoffmann, MD, MPH, Principal Investigator — Johns Hopkins University
Locations (1):
- Department of Correctional Services, Pretoria West, Pretoria, South Africa

IPD SHARING:
Plan to Share IPD: Yes
De-identified trial data will be made available one year after completion of all study activities.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: One year after completion of study activities.
Access Criteria: Contact PI

REFERENCES:
- [Derived] Mabuto T, Woznica DM, Ndini P, Moyo D, Abraham M, Hanrahan C, Charalambous S, Zack B, Baral S, Owczarzak J, Hoffmann CJ. Transitional community adherence support for people leaving incarceration in South Africa: a pragmatic, open-label, randomised controlled trial. Lancet HIV. 2024 Jan;11(1):e11-e19. doi: 10.1016/S2352-3018(23)00235-7. Epub 2023 Dec 7. PMID 38071994

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment occurred at correctional facilities between March 2019 and November 2019
Period: Overall Study
Arm/Group | Transition Community Adherence Club (TCAC) | Care as Usual (CAU)
Started | 117 | 59
Completed | 116 | 59
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Transition Community Adherence Club (TCAC) | Care as Usual (CAU) | Total
Number analyzed (Participants) | 116 | 59 | 175
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 34 [29 to 37] | 33 [29 to 36] | 33 [29 to 37]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 3 | 9
  Male | 110 | 56 | 166
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 111 | 57 | 168
  White | 4 | 1 | 5
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  South Africa | 116 | 59 | 175

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants in Care at Six Months
Description: Self-reported in TCAC or routine DoH clinical care
Time Frame: 6 months after corrections release
Measure: Count of Participants; unit: Participants
Arm/Group | Transition Community Adherence Club (TCAC) | Care as Usual (CAU)
Number analyzed (Participants) | 116 | 59
Participants | 67 | 19

2. Secondary Outcome: Proportion of Participants Verified in Care at Six Months
Description: Clinical record (electronic or paper) verified in care
Time Frame: 6 months after corrections release
Reporting Status: Not Posted

3. Secondary Outcome: Time to Linkage to HIV Care
Description: Number of days from end of intervention to first clinic visit
Time Frame: 6 months after corrections release
Reporting Status: Not Posted

4. Secondary Outcome: Proportion of Participants Linked to Care Within 90 Days of Corrections Release
Description: Self-reported in TCAC or DoH clinical care
Time Frame: 90 days after corrections release
Reporting Status: Not Posted

5. Secondary Outcome: Viral Suppression (HIV RNA <400 c/mL) at Six Months
Description: Viral load data at 6 months will be based on routinely collected viral load data (clinic records and the electronic National Health Laboratory System to determine 6 month viral load outcomes, successfully applied in prior studies) augmented by viral loads obtained by the study when 6 month viral load data are not available.
Time Frame: 6 months after corrections release
Reporting Status: Not Posted

6. Secondary Outcome: Difference in Bonding Social Capital Score at Six Months
Description: Assessed using a 12-item scale with a higher score indicating greater bonding social capital. The median scores will be compared. Range 0-48.
Time Frame: 6 months after corrections release
Reporting Status: Not Posted

7. Secondary Outcome: Difference in HIV Stigma Index Score at Six Months
Description: Assessed using 28-item Berger stigma scale with median score used per stigma construct (internalized, anticipated, experienced). Higher values indicate more stigma. Ranges: experienced 38; anticipated 6; internalized 6.
Time Frame: 6 months after corrections release
Reporting Status: Not Posted

8. Secondary Outcome: Proportion of Participants Employed or Self-employed
Description: Self-reported employment
Time Frame: 6 months after corrections release
Reporting Status: Not Posted

9. Secondary Outcome: Feasibility of Implementation of Transition Community Adherence Clubs Per Protocol (Composite Score)
Description: Feasibility of implementation will be assessed based on the proportion of participants meeting the following intervention milestones: TCAC visit, 6-month social capital questionnaire and stigma scale, and 6-month viral load ascertainment. The proportion of participants in the intervention arm who have completed all of these components with by used as a composite score (range 0-1)
Time Frame: 6 months after corrections release
Reporting Status: Not Posted

10. Secondary Outcome: Acceptability of Transition Community Adherence Clubs
Description: Qualitative outcome assessed using in-depth interviews exploring participant views on the acceptability of the transition community adherence clubs. This is a qualitative analysis based on thematic coding.
Time Frame: 6 months after corrections release
Reporting Status: Not Posted

11. Secondary Outcome: Difference in Ex-inmate Stigma Index Score at Six Months
Description: Assessed using 28-item hybrid (study specific) stigma scale with median score used per stigma construct (internalized, anticipated, experienced). Higher values indicate more stigma. Higher values indicate more stigma. Ranges: experienced 38; anticipated 6; internalized 6.
Time Frame: 6 months after corrections release
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 6 months post-corrections release
Arm/Group | Transition Community Adherence Club (TCAC) | Care as Usual (CAU)
All-Cause Mortality (participants affected / at risk) | 1/116 | 0/59
Serious Adverse Events (participants affected / at risk) | 0/116 | 0/59
Other Adverse Events (participants affected / at risk) | 0/116 | 0/59

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-04-27): https://cdn.clinicaltrials.gov/large-docs/28/NCT03340428/Prot_SAP_000.pdf
  • Informed Consent Form (2018-04-27): https://cdn.clinicaltrials.gov/large-docs/28/NCT03340428/ICF_001.pdf